CLINICAL TRIAL: NCT04809818
Title: Double-Blind, Randomized, Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of LT3001 Drug Product and Drug-Drug Interaction in Healthy Adult Subjects
Brief Title: A Study to Evaluate Safety and PK of Multiple Doses of LT3001 Drug Product and Drug-drug Interaction in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lumosa Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LT3001-105
Record Dates: First submitted 2021-03-05; First posted 2021-03-22 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin; Clopidogrel; apixaban; Dabigatran

STUDY DESIGN:
Intervention Model Description: Part A: parallel Part B: single group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A - LT3001 Drug Product (Experimental): Multiple doses of LT3001 administered by intravenous infusion
  Interventions: Drug: LT3001 drug product
- Part A - Placebo (Placebo Comparator): Multiple doses of Placebo administered by intravenous infusion
  Interventions: Drug: Placebo
- Part B - LT3001 and Aspirin (Experimental): Multiple doses of LT3001 and Aspirin administered
  Interventions: Drug: LT3001 drug product; Drug: Aspirin
- Part B - LT3001 and Clopidogrel (Experimental): Multiple doses of LT3001 and Clopidogrel administered
  Interventions: Drug: LT3001 drug product; Drug: Clopidogrel
- Part B - LT3001 and Apixaban (Experimental): Multiple doses of LT3001 and Apixaban administered
  Interventions: Drug: LT3001 drug product; Drug: Apixaban
- Part B - LT3001 and Dabigatran (Experimental): Multiple doses of LT3001 and Dabigatran administered
  Interventions: Drug: LT3001 drug product; Drug: Dabigatran

INTERVENTIONS:
Drug: LT3001 drug product — Multiple doses of LT3001 drug product administered by intravenous infusion
  Other Names: LT3001 injection
  Arms: Part A - LT3001 Drug Product; Part B - LT3001 and Apixaban; Part B - LT3001 and Aspirin; Part B - LT3001 and Clopidogrel; Part B - LT3001 and Dabigatran
Drug: Placebo — Multiple doses of Placebo administered by intravenous infusion
  Other Names: Placebo of LT3001 drug product
  Arms: Part A - Placebo
Drug: Aspirin — Loading and maintenance doses of Aspirin administered by oral
  Other Names: Aspirin tablet
  Arms: Part B - LT3001 and Aspirin
Drug: Clopidogrel — Loading and maintenance doses of Clopidogrel administered by oral
  Other Names: Clopidogrel tablet
  Arms: Part B - LT3001 and Clopidogrel
Drug: Apixaban — Multiple doses of Apixaban administered by oral
  Other Names: Eliquis®
  Arms: Part B - LT3001 and Apixaban
Drug: Dabigatran — Multiple doses of Dabigatran administered by oral
  Other Names: Pradaxa®
  Arms: Part B - LT3001 and Dabigatran

SUMMARY:
This Phase 1 study is planned to establish the clinical safety and pharmacokinetics profile of multiple dose of LT3001 drug product and to investigate drug interactions of LT3001 with potential concomitant medications in healthy subjects.

DETAILED DESCRIPTION:
This study is a two-part study. Part A is double-blind, placebo-controlled, and will examine the safety and PK profiles of multiple doses of LT3001 drug product in healthy subjects. Part B is open-label and will assess the safety and PK of LT3001 when coadministered with aspirin, clopidogrel, apixaban or dabigatran.

ELIGIBILITY:
Inclusion Criteria:

* Subject's body weight is ≥50 kg and BMI is within the range of 18 to 32
* Subject is a healthy volunteer.
* Subject's PT, aPTT, and TT are within the normal laboratory range.
* Subject is a nonsmoker

Exclusion Criteria:

* Subject has a current or recent history of regular alcohol consumption.
* Subjects who are enrolled in Part B and allergic to acetylsalicylic acid, other salicylates, clopidogrel, thienopyridines (eg, ticlopidine, prasugrel), apixaban or dabigatran.
* Part B Cohort 2 only: subjects who are poor metabolizers of clopidogrel (CYP2C19*2/*2, *2/*3, or *3/*3 genotype)
* Subject has a presence or history of coagulation abnormality.
* Subjects need to receive a surgery or clinical procedures associated with high bleeding risk.
* Subject has a history of minor bleeding episodes, eg, epistaxis, rectal bleeding, gingival bleeding.
* Subject has a history of peptic ulcer or gastrointestinal bleeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mimi Yeh, PhD, Study Director — Lumosa Phase 1 unit
Locations (1):
- Lumosa Phase 1 Unit, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A - LT3001 Drug Product: Multiple doses of LT3001 administered by intravenous infusion
  LT3001 drug product: Multiple doses of LT3001 drug product administered by intravenous infusion according to the study protocol.
- Part A - Placebo: Multiple doses of Placebo administered by intravenous infusion
  Placebo: Multiple doses of Placebo administered by intravenous infusion according to the study protocol.
- Part B - LT3001 and Aspirin: Multiple doses of LT3001 administered by intravenous infusion in combination with oral aspirin administered at loading and maintenance doses according to the study protocol.
- Part B - LT3001 and Clopidogrel: Multiple doses of LT3001 administered by intravenous infusion in combination with oral Clopidogrel administered at loading and maintenance doses according to the study protocol.
- Part B - LT3001 and Apixaban: Multiple doses of LT3001 administered by intravenous infusion in combination with oral Apixaban administered at loading and maintenance doses according to the study protocol.
- Part B - LT3001 and Dabigatran: Multiple doses of LT3001 administered by intravenous infusion in combination with oral Dabigatran administered at loading and maintenance doses according to the study protocol.
Period: Overall Study
Arm/Group | Part A - LT3001 Drug Product | Part A - Placebo | Part B - LT3001 and Aspirin | Part B - LT3001 and Clopidogrel | Part B - LT3001 and Apixaban | Part B - LT3001 and Dabigatran
Started | 12 | 4 | 13 | 12 | 12 | 12
Completed | 12 | 4 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - LT3001 Drug Product | Part A - Placebo | Part B - LT3001 and Aspirin | Part B - LT3001 and Clopidogrel | Part B - LT3001 and Apixaban | Part B - LT3001 and Dabigatran | Total
Number analyzed (Participants) | 12 | 4 | 13 | 12 | 12 | 12 | 65
Age, Categorical [Count of Participants; unit: Participants] — Population: A total of 13 subjects were enrolled in Part B Cohort 1, but only 12 subjects completed the study.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 12 | 4 | 13 | 12 | 12 | 12 | 65
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: year] | 35.5 [25 to 57] | 43.5 [22 to 54] | 45 [31 to 64] | 42.5 [28 to 61] | 45.5 [21 to 65] | 55 [30 to 62] | 42 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total of 13 subjects were enrolled in Part B cohort 1, but only 12 subjects completed the study.
  Participants
    Female | 7 | 3 | 7 | 6 | 5 | 7 | 35
    Male | 5 | 1 | 6 | 6 | 7 | 5 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 13 subjects were enrolled in Part B cohort 1, but only 12 subjects completed the study.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 6 | 2 | 0 | 0 | 2 | 1 | 11
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 1 | 1 | 5 | 5 | 2 | 3 | 17
    White | 5 | 1 | 8 | 7 | 6 | 8 | 35
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants] — Population: A total of 13 subjects were enrolled in Part B cohort 1, but only 12 subjects completed the study.
  participants
    United States | 12 | 4 | 13 | 12 | 12 | 12 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: To evaluate the safety and tolerability of LT3001 administered alone or in combination with aspirin, clopidogrel, apixaban, or dabigatran, as determined by the number and severity of adverse events collected from baseline through Day 4 post-baseline in Part A, and from baseline through Day 16 post-baseline in Part B.
Time Frame: Adverse events were assessed from baseline through Day 4 post-baseline in Part A, and from baseline through Day 16 post-baseline in Part B.
Population: Adverse events were assessed from baseline through Day 4 post-baseline in Part A, and from baseline through Day 16 post-baseline in Part B.
Measure: Number; unit: event
Arm/Group | Part A - LT3001 Drug Product | Part A - Placebo | Part B - LT3001 and Aspirin | Part B - LT3001 and Clopidogrel | Part B - LT3001 and Apixaban | Part B - LT3001 and Dabigatran
Number analyzed (Participants) | 12 | 4 | 12 | 12 | 12 | 12
event | 3 | 0 | 2 | 2 | 2 | 1

2. Secondary Outcome: Change From Baseline in Activated Partial Thromboplastin Time (APTT)
Description: Change from baseline in activated partial thromboplastin time (APTT), measured in seconds, was assessed to evaluate the safety of LT3001 administered alone or in combination with aspirin, clopidogrel, apixaban, or dabigatran from baseline up to 16 days post-dose.
Time Frame: 16 days
Population: Activated Partial Thromboplastin Time
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Part A - LT3001 Drug Product | Part A - Placebo | Part B - LT3001 and Aspirin | Part B - LT3001 and Clopidogrel | Part B - LT3001 and Apixaban | Part B - LT3001 and Dabigatran
Number analyzed (Participants) | 12 | 4 | 12 | 12 | 12 | 12
second | -0.62 (0.888) | -0.58 (0.830) | 2.62 (5.576) | 1.75 (3.349) | 0.009 (1.407) | 6.83 (4.003)

3. Secondary Outcome: Number of Participants With Prolongation in Platelet Function Test
Description: The outcome measured the number of participants with prolongation in platelet function test results following administration of LT3001 alone or in combination with aspirin, clopidogrel, apixaban, or dabigatran.
  Platelet function was assessed using collagen/epinephrine and collagen/ADP assays. Results were evaluated from baseline up to 16 days post-dose.
  Participants in the Part A placebo group did not undergo platelet function testing and were therefore not included in this outcome analysis.
Time Frame: 16 days
Population: Prolongation in collagen/epinephrine or collagen/ADP. Participants in the Part A placebo group did not undergo platelet function testing and were therefore not included in this outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - LT3001 Drug Product | Part B - LT3001 and Aspirin | Part B - LT3001 and Clopidogrel | Part B - LT3001 and Apixaban | Part B - LT3001 and Dabigatran
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Participants
  collagen/epinephrine | 0 | 1 | 1 | 0 | 0
  collagen/ADP | 1 | 5 | 4 | 0 | 2

4. Secondary Outcome: Plasma PK Parameters of LT3001 - Cmax
Description: Plasma concentrations of LT3001 and derived PK parameters up to 10 days after a single dose or multiple doses intravenous infusion of LT3001.
Time Frame: Predose and post-dose time points up to 10 days after dosing
Population: The pharmacokinetic analysis population included participants with sufficient plasma concentration data to estimate Cmax.
  Participants with missing or non-evaluable PK samples were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A - LT3001 Drug Product | Part B - LT3001 and Aspirin | Part B - LT3001 and Clopidogrel | Part B - LT3001 and Apixaban | Part B - LT3001 and Dabigatran
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 12
ng/mL | 48.86 (17.06) | 45.30 (12.31) | 43.23 (9.569) | 42.28 (15.62) | 43.96 (12.57)

5. Secondary Outcome: Plasma PK Parameters of LT3001 - Tmax
Description: as for outcome 4
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part A - LT3001 Drug Product | Part B - LT3001 and Aspirin | Part B - LT3001 and Clopidogrel | Part B - LT3001 and Apixaban | Part B - LT3001 and Dabigatran
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 12
hour | 0.22 (0.054) | 0.18 (0.073) | 0.21 (0.054) | 0.24 (0.057) | 0.21 (0.043)

6. Secondary Outcome: Plasma PK Parameters of LT3001 - AUC
Description: as for outcome 4
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A - LT3001 Drug Product | Part B - LT3001 and Aspirin | Part B - LT3001 and Clopidogrel | Part B - LT3001 and Apixaban | Part B - LT3001 and Dabigatran
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 12
h*ng/mL | 11.87 (3.364) | 9.820 (3.002) | 10.21 (2.073) | 10.32 (3.173) | 9.769 (2.558)

7. Secondary Outcome: Plasma PK Parameters of Aspirin - Cmax
Description: Plasma concentrations of Aspirin and derived PK parameters up to 8 days after multiple doses of Aspirin were administered.
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B - LT3001 and Aspirin
Number analyzed (Participants) | 6
ng/mL | 477 (362.5)

8. Secondary Outcome: Plasma PK Parameters of Aspirin - Tmax
Description: as for outcome 7
Time Frame: 8 days
Population: Participants with Plasma concentrations of Aspirin at Day 5
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part B - LT3001 and Aspirin
Number analyzed (Participants) | 6
hour | 3.7 (2.3)

9. Secondary Outcome: Plasma PK Parameters of Aspirin - AUC
Description: as for outcome 7
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part B - LT3001 and Aspirin
Number analyzed (Participants) | 6
h*ng/mL | 1709 (1251)

10. Secondary Outcome: Plasma PK Parameters of Clopidogrel - Cmax
Description: Plasma concentrations of Clopidogrel and derived PK parameters up to 10 days after multiple doses of Clopidogrel were administered.
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B - LT3001 and Clopidogrel
Number analyzed (Participants) | 12
ng/mL | 3.925 (1.991)

11. Secondary Outcome: Plasma PK Parameters of Clopidogrel - Tmax
Description: Plasma concentrations of Clopidogrel and derived PK parameters up to 10 days after multiple doses of Clopidogrel administered (alone or with LT3001).
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part B - LT3001 and Clopidogrel
Number analyzed (Participants) | 12
hour | 2.0 (1.0)

12. Secondary Outcome: Plasma PK Parameters of Clopidogrel - AUC
Description: as for outcome 10
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part B - LT3001 and Clopidogrel
Number analyzed (Participants) | 12
h*ng/mL | 8.255 (5.129)

13. Secondary Outcome: Plasma PK Parameters of Apixaban - Cmax
Description: Plasma concentrations of Apixaban and derived PK parameters up to 8 days after multiple doses of Apixaban were administered.
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B - LT3001 and Apixaban
Number analyzed (Participants) | 12
ng/mL | 188.5 (76.11)

14. Secondary Outcome: Plasma PK Parameters of Apixaban - Tmax
Description: as for outcome 13
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part B - LT3001 and Apixaban
Number analyzed (Participants) | 12
hour | 3.1 (1.5)

15. Secondary Outcome: Plasma PK Parameters of Apixaban - AUC
Description: as for outcome 13
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part B - LT3001 and Apixaban
Number analyzed (Participants) | 12
h*ng/mL | 593.8 (26.7)

16. Secondary Outcome: Plasma PK Parameters of Dabigatran - Cmax
Description: Plasma concentrations of Dabigatran and derived PK parameters up to 8 days after multiple doses of Dabigatran were administered.
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B - LT3001 and Dabigatran
Number analyzed (Participants) | 12
ng/mL | 146.1 (30.77)

17. Secondary Outcome: Plasma PK Parameters of Dabigatran - Tmax
Description: Plasma concentrations of Dabigatran and derived PK parameters up to 8 days after multiple doses of Dabigatran administered (alone or with LT3001).
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part B - LT3001 and Dabigatran
Number analyzed (Participants) | 12
hour | 4.1 (1.2)

18. Secondary Outcome: Plasma PK Parameters of Dabigatran - AUC
Description: as for outcome 17
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part B - LT3001 and Dabigatran
Number analyzed (Participants) | 12
h*ng/mL | 1807 (405.3)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from baseline through Day 4 post-baseline in Part A, and from baseline through Day 16 post-baseline in Part B.
Description: All-cause mortality, serious adverse events, and other (non-serious) adverse events were monitored during the specified adverse event reporting period. No events were observed; therefore, the number of participants at risk is reported as zero.
Arm/Group | Part A - LT3001 Drug Product | Part A - Placebo | Part B - LT3001 and Aspirin | Part B - LT3001 and Clopidogrel | Part B - LT3001 and Apixaban | Part B - LT3001 and Dabigatran
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 0/4 | 2/12 | 2/12 | 2/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - LT3001 Drug Product (N=12) | Part A - Placebo (N=4) | Part B - LT3001 and Aspirin (N=12) | Part B - LT3001 and Clopidogrel (N=12) | Part B - LT3001 and Apixaban (N=12) | Part B - LT3001 and Dabigatran (N=12)
Menstruation irregular (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracic outlet syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT04809818/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT04809818/SAP_001.pdf